CLINICAL TRIAL: NCT05633524
Title: HRR as a Novel Plasma Inflammatory Biomarker in Sjögren's Syndrome: Findings From a Case-control Study
Brief Title: HRR as a Novel Biomarker in Sjögren's Syndrome
Status: Completed | Type: Observational
Sponsor: Tianjin Eye Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: KY202226
Record Dates: First submitted 2022-11-21; First posted 2022-12-01 (Actual); Last update posted 2022-12-02 (Actual); Status verified 2022-11

CONDITIONS: Sjögren's Syndrome
MeSH Terms: conditions — Sjogren's Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 89 SS patients: The medical records were analyzed retrospectively about the 89 patients with first onset of SS (SS group)
  Interventions: Other: blood sample analysis
- 89 healthy control subjects: The medical records were analyzed retrospectively about the 89 age- and gender-matched individuals (Control group) who presented with normal control.
  Interventions: Other: blood sample analysis

INTERVENTIONS:
Other: blood sample analysis — All subjects went through a routine ocular examination, and the peripheral venous blood samples were collected and analyzed

SUMMARY:
Sjögren's syndrome (SS) is an autoimmune disorder characterized by chronic salivary and lacrimal gland dysfunction leading to dry mouth (xerostomia) and dry eye (xerophthalmia) sensation (1). Although dry mouth and dry eye are the main symptoms, the disease may influence many organs and systems. Diagnosis is made with ocular surface staining scores, anti-SS-A/SS-B auto-antibody positivity, and minor salivary gland biopsy (2). The Complete blood count (CBC) is a simple, inexpensive, accessible, and routinely used laboratory parameter that can be linked to oxidative stress, inflammation and microvascular flow resistance. Parameters include NLR and PLR values may be calculated by using CBC parameters (3). Neutrophil/lymphocyte ratio is used as an inflammatory marker in the diagnosis and prognosis of many cardiovascular diseases, malignancies, and infections (4-6). Peripheral inflammatory biomarkers of hematologic indices had been suggested by numerous studies to play a role during SS onset and progression.

DETAILED DESCRIPTION:
Sjögren's syndrome (SS) is an autoimmune disorder characterized by chronic salivary and lacrimal gland dysfunction leading to dry mouth (xerostomia) and dry eye (xerophthalmia) sensation (1). Although dry mouth and dry eye are the main symptoms, the disease may influence many organs and systems. Diagnosis is made with ocular surface staining scores, anti-SS-A/SS-B auto-antibody positivity, and minor salivary gland biopsy (2). The Complete blood count (CBC) is a simple, inexpensive, accessible, and routinely used laboratory parameter that can be linked to oxidative stress, inflammation and microvascular flow resistance. Parameters include NLR and PLR values may be calculated by using CBC parameters (3). Neutrophil/lymphocyte ratio is used as an inflammatory marker in the diagnosis and prognosis of many cardiovascular diseases, malignancies, and infections (4-6). Peripheral inflammatory biomarkers of hematologic indices had been suggested by numerous studies to play a role during SS onset and progression.

Sjögren's syndrome (SS) is a chronic autoimmune disease that primarily affects the exocrine glands, resulting in their functional impairment. In SS, lymphocytic infiltration of salivary and lacrimal glands, and deposition of several types of autoantibodies, mainly anti-SS-A (anti-Ro) and anti-SS-B (anti-La), lead to chronic inflammation, with xerostomia and keratoconjunctivitis sicca. In its primary form (pSS), SS does not involve additional connective tissue diseases. SS presents in association with other rheumatic autoimmune diseases, mainly rheumatoid arthritis (RA), systemic lupus erythematosus (SLE) and systemic sclerosis.

Obviously, a prerequisite step in answering this critical question was to depict the change of inflammatory biomarkers of hematologic indices and disease activity progression in a detailed and comprehensive manner, and actually there were several studies aimed at answering this question. Along the hematologic indices field, most of the studies agreed that RDW was critical parameter in SS activity indication.

As in most autoimmune diseases, environmental, hormonal and genetic factors are implicated in SS pathogenesis. have been shown to be a good serum marker in primary SS (pSS). All these indicated a potential linkage between systemic inflammation and the risk of SS. However, sparse evidence has been available on this association between the hematologic indices and SS. The aim of the present study, therefore, was to evaluate the association between systemic inflammation indices and SS.

ELIGIBILITY:
Inclusion Criteria:

* must meet the 2012 American College of Rheumatology classification criteria,
* without systemic diseases, such as hypertension, diabetes, cardiovascular diseases, and chronic obstructive pulmonary disease,
* without malignant tumors,
* without renal failure,
* without liver diseases,
* without anemia,
* without smoking and alcohol consumption,
* without active infection,
* without other autoimmune diseases,
* without medicine usage that could influence the blood coagulation state,
* without a history of concurrent ocular diseases or trauma,
* without any surgery within three months.

Exclusion Criteria:

* systemic diseases, such as hypertension, diabetes, cardiovascular diseases, and chronic obstructive pulmonary disease,
* malignant tumor,
* renal failure,
* liver diseases,
* anemia,
* smoking and alcohol consumption,
* active infection,
* other autoimmune diseases,
* medicine usage that could influence the blood coagulation state,
* a history of concurrent ocular diseases or trauma,
* any surgery within three months.

Ages: 45 Years to 67 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A total of 89 SS patients and 89 age- and gender-matched healthy subjects were included. Eighty-nine primary SS patients who met the 2012 American College of Rheumatology (ACR-2012) classification criteria and 89 healthy controls were enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 89 (Actual)
Dates: Start 2020-10-29 (Actual); Primary Completion 2022-11-21 (Actual); Study Completion 2022-11-21 (Actual)

PRIMARY OUTCOMES:
HRR | change from baseline at 24 months
  hemoglobin-to-red cell distribution width ratio

CONTACTS AND LOCATIONS:
Overall Officials: Yan Wang, Study Chair — Tianjin Eye Hospital and Eye Institute, Nankai University Affiliated Eye Hospital
Locations (1):
- Tianjin Eye Hospital, Tianjin, Tianjin Municipality, China

REFERENCES:
- [Result] Psianou K, Panagoulias I, Papanastasiou AD, de Lastic AL, Rodi M, Spantidea PI, Degn SE, Georgiou P, Mouzaki A. Clinical and immunological parameters of Sjogren's syndrome. Autoimmun Rev. 2018 Oct;17(10):1053-1064. doi: 10.1016/j.autrev.2018.05.005. Epub 2018 Aug 10. PMID 30103041
- [Result] Yildiz F, Gokmen O. Haematologic indices and disease activity index in primary Sjogren's syndrome. Int J Clin Pract. 2021 Mar;75(3):e13992. doi: 10.1111/ijcp.13992. Epub 2021 Jan 19. PMID 33405348
- [Result] Hu ZD, Sun Y, Guo J, Huang YL, Qin BD, Gao Q, Qin Q, Deng AM, Zhong RQ. Red blood cell distribution width and neutrophil/lymphocyte ratio are positively correlated with disease activity in primary Sjogren's syndrome. Clin Biochem. 2014 Dec;47(18):287-90. doi: 10.1016/j.clinbiochem.2014.08.022. Epub 2014 Sep 7. PMID 25204965